CLINICAL TRIAL: NCT04008823
Title: Study of Influenza Virus Infection in Children Hospitalized in Spain in Two Consecutive Influenza Seasons. Analysis of Direct Medical Costs
Brief Title: Study of Influenza Virus Infection in Children Hospitalized in Spain in Two Consecutive Influenza Seasons
Acronym: HOSPIGRIP
Status: Completed | Type: Observational
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HOSPIGRIP
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Influenza Virus Infection
MeSH Terms: interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective and observational epidemiological study, by review of clinical histories, — Retrospective and observational epidemiological study, by review of clinical histories,

SUMMARY:
This is an epidemiological, retrospective and observational study, by reviewing clinical histories, of children hospitalized for influenza virus infection, their comorbidities and the treatments that have been performed

DETAILED DESCRIPTION:
A better knowledge in our environment of the characteristics of the Influenza virus infection in the pediatric age, the clinical aspects, risk factors, the evolutionary and prognostic aspects, of morbidity and the direct medical costs, can allow a better management of the disease and a greater awareness of the importance of vaccination against influenza in the healthy child

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls under 15 years of age.
* With a clinical diagnosis of influenza virus infection.
* With infection by influenza virus confirmed microbiologically.
* Hospitalized more than 24 hours

Exclusion Criteria:

* Age equal to or greater than 15 years.
* That the clinical diagnosis is not influenza virus infection.
* Influenza virus not confirmed by microbiological diagnosis.
* Not hospitalized or hospitalized for less than 24 hours.

Age Groups: Child, Adult, Older Adult
Study Population: the population under study is children under 15 years of age, hospitalized for infection with influenza virus confirmed microbiologically during two consecutive seasons (September 15, 2014 to June 30, 2015) (September 15, 2015 to June 30, 2015). 2016).
Sampling Method: Non-Probability Sample
Enrollment: 907 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
To study the rate of hospitalizations for influenza virus infection in children under 15 years of age in third level hospitals in Spain. | 2014-2016
  Number of hospitalizations in children under 15 years old due to influenza virus infection

SECONDARY OUTCOMES:
Hospitalization rate by age groups (0-6 months, 6 months to 24 months, 2 to 6 years, 6 to 10 years and 10 to 15 years of age | 2014-2016
Demographic characteristics of hospitalizations for influenza in children | 2014-2016
  Age, sex, weight
Complications associated with influenza infection. | 2014-2016
Related morbidity | 2014-2016
Estimation of direct costs | 2014-2016
  * Income costs and prescribed medication.
  * Test costs.
  * Bed and UCIP costs.
  * Costs previous visits (to hospitalization) to the emergency room
Epidemiological characteristics of hospitalizations for influenza in children | 2014-2016
  Presence or absence of seasonal influenza vaccination.
Clinical characteristics of hospitalizations for influenza in children | 2014-2016
  * Presence / absence in microbiological analysis of influenza virus.
  * Coinfections.
  * Presence or absence of complications during hospitalization.
  * Variables of clinical evolution.
  * Analytical variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Iis Biodonostia, San Sebastián, Guipuzcoa, Spain

IPD SHARING:
Plan to Share IPD: No